CLINICAL TRIAL: NCT05450965
Title: A Phase 2 Study of PLK1 Inhibitor, Onvansertib, in Relapsed Small Cell Lung Cancer
Brief Title: Study of PLK1 Inhibitor, Onvansertib, in Relapsed Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Cardiff Oncology (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2412GCCC ; HP-00109457; R01CA273216-01 (NIH)
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Carcinoma
Keywords: Lung Cancer; Onvansertib; Polo-like Kinase; PLK1; Salvage Therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — onvansertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Treatment Arm (Experimental): Onvansertib
  Interventions: Drug: Onvansertib

INTERVENTIONS:
Drug: Onvansertib — Onvansertib at a dose of 15 mg/m2 orally on Days 1-14 of a 21-day cycle. Treatment will continue until disease progression or intolerable toxicity.

SUMMARY:
This phase II clinical trial will study the safety and efficacy of onvansertib to treat patients with small cell lung cancer (SCLC) who have either not responded to or are unable to tolerate chemotherapy. Onvansertib is a drug that inhibits polo-like kinase 1 (PLK-1), an enzyme that is over-expressed in many cancer cells and is involved in cellular repair.

DETAILED DESCRIPTION:
This is a single arm, two stage, phase II study of onvansertib in patients with relapsed SCLC who have received not more than 2 lines of prior therapies. The study will enroll 15 patients in stage I. Enrolment into stage II will occur if two or more patients achieve objective response. Subsequent enrolment into stage II will be by biomarker selection if the stage I accrual supports any of the three preliminarily nominated biomarkers i.e., TP53 mutation type, SCLC-Y or MYC expression. In order to establish the safety and tolerability of onvansertib at the dose of 15 mg/m2 on D1-D14 of a 21-day cycle, the first 6 participants will be closely monitored as a safety a run-in. Full safety evaluation will be conducted after all 6 patients have completed at least 1 cycle of therapy. A lower dose of onvansertib will be considered, and schedule of onvansertib as per the planned dose modification strategy, if during the safety run-in there are any deaths not clearly attributable to the underlying disease or extraneous causes or for Grade 4 hematologic or non-hematologic adverse events (AEs) occurring in 2 or more patients. In the event that a dose de-escalation is necessary following the initial safety run-in cohort, the run-in procedure will be repeated for the reduced dose level as described above. The study will continue to enroll to stage I at the dose established to be safe from the safety run-in cohort. Patients treated at the established dose in the safety run-in phase will count toward the total stage I accrual goal of 15 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed small cell lung cancer
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 8for the evaluation of measurable disease.
3. Patient must have failed or found to be intolerant of standard frontline platinum-based regimens and not more than two lines of cytotoxic chemotherapy treatment in total for extensive stage disease. Maintenance immunotherapy counts as part of the frontline therapy, while prior chemotherapy for limited stage disease will not count toward this total if completed more than 12 months before initiation of protocol therapy. Retreatment with the original chemotherapy regimen for sensitive relapsed SCLC counts as a separate line of treatment.
4. Adult patients with age >18 years. Because no dosing or adverse event data are currently available on the use of arsenic trioxide in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
5. Ability to tolerate oral medicine
6. ECOG performance status ≤2
7. Patients must have normal organ and marrow function as pre-defined
8. Negative serum pregnancy test within 48 hours before starting study treatment in women with childbearing potential
9. Women of child-bearing potential and men must agree to use adequate contraception.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

1. Treatment with chemotherapy (within 4 weeks; 6 weeks for nitrosoureas or mitomycin C); radiotherapy or biologic agents (within 2 weeks) prior to first dose of onvansertib or those persistent, clinically significant, grade ≥2 adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents (Use of conventional external beam radiation therapy will be allowed during protocol therapy solely for palliation of localized painful lesions or bone lesions at risk of fracture provided the radiation field does not encompass any selected target lesions required for assessment).
3. Patients with uncontrolled symptomatic brain metastases. Subjects with a history of central nervous system (CNS) metastases must have documentation of stable brain imaging after completion of definitive treatment and prior to first dose of Study Drug. Patients must be off or on a stable dose of corticosteroids (not more than 10mg prednisone or equivalent). Definitive treatment may include surgical resection, whole brain irradiation, and/or stereotactic radiation therapy.
4. Patients with active GI disorders likely to impair the absorption of oral medications
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to onvansertib.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patient with untreated or active HBV, HCV and HIV are ineligible. Patients on stable doses of antiretroviral for at least six months and undetectable viral load will be enrolled with prior approval of the study sponsor. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
8. Patients who require ongoing treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug.
9. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
10. Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 42 months (cohort)
  The proportion of patients having either a complete response (CR) or partial response (PR) (as best response), per RECIST 1.1. Complete Response (CR): Disappearance of all target lesions. For non-target lesions, CR is the disappearance of all non-target lesions and normalization of tumor marker level. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 3.5 years
  The number of patients incurring specific Adverse Events or Serious Adverse Events that occur from first day of treatment, considered to be possibly, probably or definitely related to study treatment, per Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Patients experiencing multiple AEs of the same type will be reported by only the most severe grade.
Progression-free survival (PFS) | Up to 3.5 years
  The median number of months from start of treatment to time of disease progression or death (from any cause), whichever occurs first. Progressive Disease (PD) as defined by RECIST v1.1 for target lesions: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Overall survival (OS) | Up to 3.5 years
  The median number of months from start of treatment to time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, MD, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang G, Pannucci A, Ivanov AA, Switchenko J, Sun SY, Sica GL, Liu Z, Huang Y, Schmitz JC, Owonikoko TK. Polo-like Kinase 1 Inhibitors Demonstrate In Vitro and In Vivo Efficacy in Preclinical Models of Small Cell Lung Cancer. Cancers (Basel). 2025 Jan 28;17(3):446. doi: 10.3390/cancers17030446. PMID 39941812